CLINICAL TRIAL: NCT04702633
Title: Non-invasive Isolation and Characterization of Prostate Tumor Cells for Prostate Cancer Diagnosis
Brief Title: Immuno-molecular Approaches for Non-invasive Diagnosis of Prostate Cancer
Acronym: PROSTA-PAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Rarecells Diagnostics SAS (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201309
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Liquid biopsy; Biological samples; Non-invasive diagnosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples (blood, plasma, urines) and paraffin-embedded tissue cuts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed diagnosis group: Patients with a diagnosis of prostate cancer (metastatic or advanced) before prostatectomy.
  Interventions: Other: Results obtained by biopsy and MRI results.; Other: Clinical data
- Pre-diagnosis group: Patients undergoing prostate biopsy in the context of prostate cancer diagnosis: PSA increases, and / or abnormal digital rectal examination (DRE) and / or an MRI detected signal.
  Interventions: Other: Results obtained by biopsy and MRI results.; Other: Clinical data

INTERVENTIONS:
Other: Results obtained by biopsy and MRI results. — Results obtained by biopsy and MRI results.
Other: Clinical data — Clinical data

SUMMARY:
The purpose of this study is to isolate and characterize tumor cells non-invasively from biological samples in patients with prostate cancer and demonstrate the ability to identify the presence and number of tumor cells before prostate biopsy.

DETAILED DESCRIPTION:
Prostate cancer is one of the most frequently diagnosed cancers and a leading cause of cancer death in men worldwide. Existing methods of diagnosis and monitoring of prostate cancer are inadequate due to their invasiveness, inaccuracy, cost, access uneven, etc., making difficult the diagnosis and patient's follow up. New techniques and methods are necessary to improve diagnosis.

Biological liquids might represent an attractive target to isolate prostate tumour cells for these purposes. In recent years, several studies have been carried out with the aim of reducing and / or avoiding the limits of sensitivity and specificity of current methods of screening for prostate cancer and thus obtain new biomarkers for the diagnosis and / or non-invasive monitoring.

However, due to technical and technological difficulties few studies have been performed to investigate the non-invasive isolation and direct analysis of tumour cells. Our project is therefore an innovative project which aims to study a new approach for the early diagnosis of prostate cancer, with better sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of localized or metastatic prostate cancer.
* No prior or other oncological treatment.
* Patients undergoing prostate biopsy in the context of prostate cancer diagnosis.
* Patients with an elevation of PSA (Prostate Specific Antigen), an abnormality on the rectal examination and / or an MRI signal motivating a prostate biopsy,
* Patients informed and not opposed to participating in the research

Exclusion Criteria:

* Patients not affiliated with French social security.
* Patients unable to understand the protocol.
* Patients diagnosed with another type of cancer within the past 5 years.
* Patients prostatectomized and/or treated for prostate cancer.
* Patients who wear a bladder catheter
* Patients under guardianship or curatorship
* Patients under AME

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting the urology department of Cochin Hospital with an indication for prostate biopsy or as part of the monitoring of prostate cancer may be included.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Presence and number of prostate tumour cells in biological samples | One month after biopsy or until the histological diagnosis will be obtained
  Cell enrichment will be carried out using the ISET® (Isolation by SizE of Tumor/Trophoblastic cells) technology. Identification will be performed by different spectroscopic and/or immune-molecular and/or cytological approaches

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia PATERLINI-BRECHOT, MD, PhD, Study Chair — INSERM and Rarecells Diagnostics
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No